CLINICAL TRIAL: NCT02819479
Title: Low-dose Intra-arterial Bevacizumab for Edema and Radiation Necrosis Therapeutic Intervention (LIBERTI)
Acronym: LIBERTI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norton Healthcare (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Principal Investigator, Shervin Dashti, MD, Principal Investigator, Norton Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-N0229
Record Dates: First submitted 2016-05-09; First posted 2016-06-30 (Estimated); Results first posted 2021-06-28 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Radiation Necrosis
Keywords: Radiation necrosis; Radiation adverse event; Intra-arterial chemotherapy; Bevacizumab; Blood brain barrier disruption; Blood brain barrier breakdown; Arteriovenous malformation; Stereotactic radiosurgery
MeSH Terms: conditions — Arteriovenous Malformations | interventions — Mannitol; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low-dose Intra-arterial Bevacizumab (Experimental): A single intra-arterial targeted dose of 2.5 mg/kg bevacizumab will be administered after osmotic blood-brain-barrier disruption with intra-arterial 25% mannitol at rate of 4-12 ml/sec for 30 seconds.
  Interventions: Drug: 25% Mannitol; Drug: Low-dose Intra-arterial Bevacizumab

INTERVENTIONS:
Drug: 25% Mannitol — Route of administration:
  In this study, the first step of the treatment will be performing osmotic blood-brain-barrier disruption with administration of intra-arterial 25% Mannitol into the appropriate cervical artery.
Drug: Low-dose Intra-arterial Bevacizumab — Route of administration:
  In this study, the second step of the treatment will be administering intra-arterial targeted bevacizumab into the appropriate cervical artery.
  Other Names: Avastin

SUMMARY:
To assess the overall safety and efficacy of intra-arterial (IA) bevacizumab for the treatment of radiation necrosis. A single 2.5 mg/kg dose of bevacizumab will be given intra-arterially after osmotic blood-brain-barrier disruption.

DETAILED DESCRIPTION:
BACKGROUND Radiation Necrosis: Stereotactic radiosurgery has become integral in treatment of brain tumors and arteriovenous malformations (AVM). In up to 10% of cases, this can lead to radiation necrosis (RN) with significant surrounding vasogenic edema and mass effect. Medical treatment for RN includes steroids, vitamin E, pentoxiphylline, and hyperbaric oxygen. Up to 20% of cases however, are medically refractory and experience progressive neurological decline and disabling headaches.

Surgical resection and laser interstitial thermal therapy (LITT) are sometimes used for treatment of medically refractory radiation necrosis. These invasive options carry risks of serious complications such as infection, seizures, neurological deficits, and hemorrhage, and may have a failure rate as high as 39% in patients with radiation necrosis of the brain.

Bevacizumab: Bevacizumab (Avastin, Genentech BioOncology, South San Francisco, CA) is a recombinant humanized version of a murine anti-human vascular endothelial growth factor (VEGF) monoclonal antibody. Recently, bevacizumab was shown in a small randomized controlled trial (n=14) to be effective in treatment of refractory radiation necrosis after radiation therapy in brain tumors1. Patients received 7.5 mg/kg IV-Bevacizumab every 3 weeks for 4 cycles. All patients receiving Bevacizumab and none of the patients receiving placebo had significant clinical and radiographic improvement.

PRE-CLINICAL DATA Role of vascular endothelial growth factor (VEGF) in radiation necrosis VEGF has been implicated in the pathophysiology of radiation necrosis. Reactive astrocytes immediately surrounding the necrotic core in RN are strongly VEGF-positive by immunohistochemistry. It is postulated that radiation causes microvascular injury leading to hypoxia. Hypoxia-induced VEGF up-regulation then drives an increase in vascular permeability, leading to the extensive vasogenic edema seen in RN. Bevacizumab binds circulating VEGF receptors with high specificity, blocking the down-stream signaling cascade.

CLINICAL DATA:

Bevacizumab was originally developed and tested as an anti-angiogenic treatment for various solid tumors. More recently, IV-Bevacizumab was shown in a small, randomized controlled trial (n=14) to be very effective in treatment of refractory radiation necrosis after radiation therapy in brain tumors1. Patients received 7.5 mg/kg IV-Bevacizumab every 3 weeks for 4 cycles. All patients receiving Bevacizumab and none of the patients receiving placebo had significant clinical and radiographic improvement. This improvement was durable at 10 months in 8 of 11 patients (4 patients crossed over from the control group). There was however, a very high rate of adverse events (60%), and major adverse events (30%). Major adverse events included venous sinus thrombosis, pulmonary embolus, and aspiration pneumonia.

The investigators of the present study recently published a case series of two pediatric patients with highly symptomatic steroid refractory radiation necrosis in the brain after stereotactic radiosurgery for treatment of cerebral arteriovenous malformations3. Both patients were refractory to all accepted medical therapies. Both were steroid dependent for a prolonged period and severely cushingoid. Both had suffered a significant decline in quality of life with severe headache and needed to withdraw from school. In both instances, the patients made a remarkable progressive clinical and radiographic improvement after receiving a single 2.5 mg/kg dose of intra-arterial bevacizumab, which was durable one-year later. To increase bevacizumab penetration into the brain, the investigators used intra-arterial Mannitol to disrupt the blood-brain barrier immediately prior to targeted intra-arterial drug administration.

RATIONALE:

RATIONALE: CURRENT IV BEVACIZUMAB REGIMEN FOR RADIATION NECROSIS AND ITS ASSOCIATED MORBIDITY:

Current IV-bevacizumab regimens use a dose of 7.5 mg/kg every 3 weeks for 4 cycles. There are significant known side effects of bevacizumab including gastrointestinal perforation, deep venous thrombosis, venous sinus thrombosis, pulmonary embolus, intracranial hemorrhage, wound dehiscence, and severe hypertension. These complications are common to the anti-angiogenic class of drugs and reflect systemic exposure to bevacizumab. In our initial clinical experience, the investigators utilized a combination of intra-arterial (IA) route of delivery and BBB disruption to reduce bevacizumab dose while maintaining efficacy. This is supported by the durable clinical and radiographic response in our patients after a single 2.5 mg/kg dose of bevacizumab. The investigators believed that this approach would reduce the incidence of serious systemic toxicities compared to the IV-bevacizumab regimens (7.5-15 mg/kg every 2-3 weeks for several weeks to months).

There are multiple recent reports of patients with radiation necrosis who improved with IV-bevacizumab, only to relapse months later. In fact 3/11 patients in the randomized controlled trial discussed above required repeat treatment with IV-bevacizumab because of RN symptom progression1. In contrast, the two patients in our series who received IA-bevacizumab continue to show progressive clinical and radiographic improvement more than one year later. The investigators believe that the increased penetration of bevacizumab into the brain because of the intra-arterial administration after blood-brain barrier disruption results in binding of virtually all VEGF molecules. The fact that the results are durable and progressively improving suggests that massive blocking of VEGF activity could have stopped a positive feedback loop of inflammation. Therefore, IA-bevacizumab may result in more effective and durable control of radiation necrosis compared to traditional IV-bevacizumab treatment.

RATIONALE: INTRA-ARTERIAL (IA) ROUTE OF BEVACIZUMAB ADMINISTRATION SIGNIFICANTLY INCREASES DRUG DELIVERY TO THE BRAIN:

IA-therapy decreases volume dilution of the drug in the circulation and reduces first-pass degradation via proteolytic catabolism, resulting in higher drug delivery to target brain tissue. Super-selective IA-injection of 99mTc-HMPAO (Ceretec®) into human cerebral arteries achieves a concentration of radiotracer in brain tissue 50 times higher than with IV injection. In clinical studies of cerebral chemotherapy, the concentration delivered to the tumor by using intra-arterial injection versus intravenous administration of chemotherapeutic agents was five times higher with hydrosoluble drugs and up to 50 times higher with liposoluble drugs. The investigators will infuse bevacizumab in the artery that supplies the territory affected by RN, such as cervical internal carotid artery and/or cervical vertebral artery.

RATIONALE: BLOOD-BRAIN-BARRIER BREAKDOWN PRIOR TO INTRA-ARTERIAL THERAPY FURTHER ENHANCES DRUG DELIVERY TO THE BRAIN:

The blood-brain-barrier is a selective permeability barrier that block entry of many drugs into the brain. Bevacizumab is a monoclonal antibody with a high molecular weight (149 kDa). There is convincing evidence in the literature that the concentration in the brain of high molecular weight molecules can be significantly increased after osmotic BBB disruption. Several tumor clinical trials have shown that localization of monoclonal antibodies to the brain is poor without BBB disruption (0.0006%-0.0043% of the injected dose/g of tumor). There is also evidence of a 20-fold increase in permeability to immunoreactive IgM Mab with BBB disruption in rats. The investigators believe that using blood-brain-barrier disruption significantly increases delivery of Bevacizumab to the affected brain. The investigators will use the protocol described by Neuwelt and colleagues, using infusion of 25% Mannitol over 30 seconds. This protocol has been shown to temporarily disrupt the blood brain barrier, peaking at 15 minutes and dissipating in 4 hours. IA-chemotherapy following BBBD has been shown to be feasible and safe across multiple centers with low incidence of complications27. The efficacy and safety profile was reproducible across multiple centers. In fact, safety of this protocol has been established in more than 6000 patients treated worldwide with BBBD for intra-arterial chemotherapy infusion. The main possible complication is seizure, which occurs in <6% of cases. It is important to note that these seizures generally occurred in patients with widespread malignant pathology such as Glioblastoma and CNS lymphoma who were treated with very toxic chemotherapy agents immediately after BBBD. Recent refinements to the osmotic BBBD protocol have incorporated the use of general anesthesia, as well as prophylaxis with an anti-epileptic agent and Valium to reduce seizure threshold and the chance of seizures.

SAFETY OF CEREBRAL INTRA-ARTERIAL BEVACIZUMAB TREATMENT:

Safety of IA-Bevacizumab treatment after hyperosmotic BBBD was recently established in a series of malignant glioma patients. This was done through super-selective injection of intracranial tumor arterial pedicles for purpose of anti-tumor effects. Dose-escalation was performed from 2 mg/kg to 15 mg/kg without reaching maximal tolerated dose. There was a significant decrease in the contrast enhancing and FLAIR signal characteristics of the tumor and surrounding brain at one month after treatment. Overall toxicity for this cohort was comparable to previous reports for IV Bevacizumab therapy. Specifically, hyperosmotic BBB-breakdown followed by IA-Bevacizumab administration did not cause any direct neurotoxicity; there were no cases of intracranial hemorrhage. Multiple other reports of BBBD followed by intra-arterial bevacizumab treatment for other pathologies such as vestibular schwannoma, ependymoma, and malignant brainstem glioma have also demonstrated good safety profile with no obvious neurotoxicity.

TREATMENT PLAN:

VASCULAR ACCESS, CEREBRAL ANGIOGRAM, AND OSMOTIC BLOOD-BRAIN-BARRIER DISRUPTION:

The investigators will use the protocol described by Neuwelt and colleagues, using infusion of 25% Mannitol over 30 seconds. The safety of this protocol has been established in more than 6000 patients treated worldwide with BBBD for intra-arterial chemotherapy infusion.

The patients are to be premedicated with 6 mg Dexamethasone and 1000 mg Keppra. General endotracheal anesthesia will be induced. The femoral artery will be accessed using the Seldinger technique. A 5-French diagnostic catheter will be used to catheterize the cervical internal carotid artery ipsilateral to the area of radiation necrosis. Baseline internal carotid angiogram will be performed.

The anesthesiologist will be instructed to maintain SBP >120 or at pre-operative baseline, whichever value is higher. This is important for efficient bulk flow of drug through the blood brain barrier opening. The catheter is positioned at C1-2 level in the cervical internal carotid artery and C6-7 for a vertebral artery infusion. Optimal rate of Mannitol infusion will be determined by performing injection of contrast at 4 ml/sec for 3 seconds into vessel. If there is no reflux of contrast into the external carotid artery, the injection rate injection will be increased by 2 ml/sec to maximum of 12 ml/sec. The lowest rate at which there is reflux into the external carotid artery will be chosen (the rate to just exceed cerebral blood flow.

Next, 5 mg IV Valium and 0.2 mg IV Atropine are to be administered. Warm (37 degrees Co) 25% Mannitol is filtered through a 5-micron filter, and then infused into the ipsilateral cervical carotid artery at the rate determined above for a total of 30 seconds.

INTRA-ARTERIAL BEVACIZUMAB ADMINISTRATION:

Test injection of contrast will be done in the artery. If there is any evidence of catheter-induced vasospasm, the catheter may be withdrawn more proximally within the artery. Repeat test injection of contrast will be done to document resolution of vasospasm. Within 5 minutes of Mannitol infusion, 2.5 mg/kg bevacizumab in a volume of 100 ml will be administered into the artery over 10 minutes. Repeat angiogram will be performed to document BBBD, as well as to rule out thromboembolic phenomenon.

ELIGIBILITY:
Inclusion Criteria:

Patients must have radiation necrosis based on radiographic evidence defined as:

* Increased T1 contrast enhancement in the radiated area with central hypointensity
* Increased surrounding vasogenic edema on FLAIR MRI images
* The underlying lesion prompting the radiation can include: Benign lesions such as AVM, Meningioma, schwannoma, trigeminal neuralgia: No biopsy is necessary
* Radiation necrosis must be symptomatic, including either severe headache, seizures, or neurological deficits.
* Radiation necrosis must be refractory to steroid treatment; defined as failing a 3-week steroid regiment or not tolerating steroids because of side effects. Beyond 3 weeks, the side effects of steroid therapy worsen rapidly. The patient may receive other therapies such as Vitamine E, Pentoxyfylline, and hyperbaric oxygen during the trial.

Other inclusion criteria include:

* Age >18 years.
* Ability to understand and the willingness to sign a written informed consent document.
* Both men and women and members of all races and ethnic groups are eligible for this trial.
* Karnofsky Performance Status > or = 70%.
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined below:

leukocytes greater than equal to1,500/mcL platelets greater than equal to 85,000/mcL creatinine less than equal to 1.8 mg/dl

•Birth Control: The effects of Bevacizumab on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Women of childbearing age will have a urine pregnancy test immediately before each IA Bevacizumab treatment.

Exclusion Criteria:

* Patients may not be started on any other investigational agents during the course of this trial. They may however continue previous medical regiments aimed for treatment of radiation necrosis. These include steroids, vitamin E, pentoxiphylline, and hyperbaric oxygen. We feel that these treatments are generally ineffectual and would not confound the results.
* Malignant brain tumor
* Concomitant use of anticoagulation agents including Coumadin, anticoagulation dose Lovenox or Arixtra. Aspirin is acceptable.
* Active bleeding or pathological condition that carries high risk of bleeding.
* Abdominal fistula, abscess, or gastrointestinal tract perforation 28 days of study entry.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any major surgery in the prior 4 weeks. Also any major surgery expected to be performed in the ensuing 4 weeks after treatment.
* Pregnant women are excluded from this study because Bevacizumab is expected to disrupt angiogenesis during pregnancy with the potential for teratogenic or abortive effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Bevacizumab, breastfeeding should be discontinued if the mother is treated with Bevacizumab.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shervin R Dashti, MD,PhD, Principal Investigator — Norton Healthcare; Justin Fraser, MD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Norton Brownsboro Hospital, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dashti SR, Kadner RJ, Folley BS, Sheehan JP, Han DY, Kryscio RJ, Carter MB, Shields LBE, Plato BM, La Rocca RV, Spalding AC, Yao TL, Fraser JF. Single low-dose targeted bevacizumab infusion in adult patients with steroid-refractory radiation necrosis of the brain: a phase II open-label prospective clinical trial. J Neurosurg. 2022 Apr 15;137(6):1676-1686. doi: 10.3171/2022.2.JNS212006. Print 2022 Dec 1. PMID 35426830

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults recruited from outpatient medical clinics at 2 academic medical centers (5 subjects per center) between Nov 2016 and Jan 2018. Enrollment was closed once 10 adult subjects were enrolled.
Pre-assignment Details: This was a single-arm study. There was no wash out or run-in period after enrollment. There was no assignment to groups.
Groups:
- Low-dose Intra-arterial Bevacizumab: A single intra-arterial dose of 2.5 mg/kg bevacizumab will be administered after osmotic blood-brain-barrier disruption with intra-arterial 25% mannitol at rate of 4-12 ml/sec for 30 seconds.
  25% Mannitol: Route of administration: In this study, the first step of the treatment will be performing osmotic blood-brain-barrier disruption with administration of intra-arterial 25% Mannitol into the appropriate cervical artery.
  Low-dose Intra-arterial Bevacizumab: Route of administration:
  In this study, the second step of the treatment will be administering intra-arterial bevacizumab into the appropriate cervical artery.
Period: Overall Study
Arm/Group | Low-dose Intra-arterial Bevacizumab
Started | 10
Completed | 8 (2 subjects experienced recurrence of radiation necrosis requiring intervention at approx. month 11.)
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Low-dose Intra-arterial Avastin (Bevacizumab): A single intra-arterial dose of 2.5 mg/kg bevacizumab will be administered after osmotic blood-brain-barrier disruption with intra-arterial 25% mannitol at rate of 4-12 ml/sec for 30 seconds.
  25% Mannitol: Route of administration: In this study, the first step of the treatment will be performing osmotic blood-brain-barrier disruption with administration of intra-arterial 25% Mannitol into the appropriate cervical artery.
  Low-dose Intra-arterial Bevacizumab: Route of administration:
  In this study, the second step of the treatment will be administering intra-arterial bevacizumab into the appropriate cervical artery.
Arm/Group | Low-dose Intra-arterial Avastin (Bevacizumab)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment, years
  years | 35.1 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
MRI of Brain: volume of radiation necrosis [Mean (Standard Deviation); unit: cubic centimeters, or cm^3] | 14.5 (12.1)
MRI of Brain: volume of edema [Mean (Standard Deviation); unit: cubic centimeters, or cm^3] | 86.8 (95.9)
Headache severity via Migraine Disability Assessment (MIDAS) TOTAL SCORE [Mean (Standard Deviation); unit: units on a scale from 0 to 450] — MIDAS (Migraine Disability Assessment) is a 7-item tool that measures how severely headaches prevented or interfered with normal activity over the past 3 months. For each item 1 through 5 the min score=0 days, max score=90 days. The MIDAS TOTAL SCORE sums items 1 - 5 only. TOTAL SCORE of 0-5 indicates little or no disability. Total Score of 6-10 indicates mild disability. Total Score of 11-20 indicates moderate disability. Total score of 21+ indicates severe disability. Theoretical Max Total Score is 450 days.
  units on a scale from 0 to 450 | 81.7 (110.1)
DAYS of Headache via Migraine Disability Assessment (MIDAS) [Mean (Standard Deviation); unit: Days of headache over past 3 months] — MIDAS (Migraine Disability Assessment) questionnaire is a 7-item tool that measures how severely headaches prevented or interfered with normal activity over the past 3 months. MIDAS DAYS of HEADACHE is Item 6 of the questionnaire which sums total number of days the patient had headache symptoms over the past 3 months regardless of headache severity or resultant disability. Min score of 0 days is the best possible score. Max Score of 90 days is worse possible score, meaning the patient experienced headache pain every day over past 3 months.
  Days of headache over past 3 months | 33.3 (29.8)
Headache PAIN LEVEL via Migraine Disability Assessment (MIDAS) [Mean (Standard Deviation); unit: units on a scale from 0 to 10] — MIDAS (Migraine Disability Assessment) is a 7-item tool that measures how severely headaches prevented or interfered with normal activity over the past 3 months. Item 7 rates the 3-month average headache PAIN LEVEL on scale from 0 to 10 where 0 = no pain at all, and 10 = pain as bad as it can be.
  units on a scale from 0 to 10 | 6.9 (2.2)
Headache severity via Headache Impact Test (HIT-6) [Mean (Standard Deviation); unit: units on a scale from 36 - 78] — The Headache Impact Test-6 is a tool used to measure the impact headaches have on a patient's ability to function in their normal daily life. This 6-item questionnaire was designed to help patients describe and communicate the way they feel and what they cannot do because of their headaches. For each item, patients must select one answer: never, rarely, sometimes, very often, or always. Scores range from min of 36 indicating minimum headache impact, to a max of 78 indicating worst possible headache impact. A score of 60 or more indicates headaches having a very severe impact on daily life.
  units on a scale from 36 - 78 | 62.4 (7.5)
Cumulative Days of Steroid use during 12 months Pre-Bevacizumab [Median (Inter-Quartile Range); unit: Days] — Total cumulative days of steroid usage were compared between the 12 months prior to and the 12 months immediately following targeted IA-bevacizumab. Days of steroid usage was tabulated via medical history and chart review at the baseline visit, and post-treatment on days 0 and 1, week 6, and months 3, 6, 9 and 12. Excluding topical steroid preparations, all days of enteral or parenteral steroid intake of any dose were included in the cumulative summation.
  Days | 52.5 [0 to 100]
Karnofsky Performance Status Scale [Mean (Standard Deviation); unit: % on Karnofsky scale] — The Karnofsky Performance Status Scale allows patients to be classified as to their functional impairment. The lower the score, the worse the survival for most serious illnesses. Scores range from 0% to 100% where 100%=Normal with no complaints, no evidence of disease. 90%=Able to carry on normal activity; minor signs or symptoms of disease. 80%=Normal activity with effort; some signs or symptoms of disease. 70% = cares for self; unable to carry on normal activity or to do active work. 60%=Requires occasional assistance, but is able to care for most of his personal needs and 0%=Dead.
  % on Karnofsky scale | 79.0 (9.9)
Digits Forward via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically adjusted, normalized battery of tests which measure neurocognitive function. The Digits Forward module generates T scores which indicate the degree to which immediate auditory attention is higher or lower than that of healthy demographically matched individuals in the normative sample. T-score of 50 is the mean and is considered normal. Scores significantly below 40 indicate decreased auditory attention. Scores significantly above 60 indicate better auditory attention than healthy demographically matched persons.
  T score with Mean=50, SD=10 | 41.1 (11.8)
Digits Backward via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically adjusted, normalized battery of tests which measure neurocognitive function. The Digits Backward module generates T scores which indicate the degree to which auditory working memory is stronger or weaker than that of a healthy demographically matched individual in the normative sample. T-score of 50 is equal to the mean and is considered normal. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 44.9 (8.3)
Numbers and Letters Speed via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically adjusted normalized battery of tests which measure neurocognitive function. Numbers & Letters Speed module is an excellent general indicator of speed and efficiency of information processing. T scores indicate the degree to which info processing speed differs from that of healthy demographically matched individuals. T-scores of 40-60 are within 1 SD of the mean (50) and are considered normal. Scores below 40 indicate decreased processing speed. Scores above 60 indicate more rapid processing speed.
  T score with Mean=50, SD=10 | 38.2 (10.7)
Numbers and Letters Errors via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. Numbers & Letters ERRORS module measures the extent of errorful processing. Errorful processing is considered "inefficient". T scores indicate the degree to which processing efficiency differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 44.6 (3.8)
Numbers and Letters Efficiency via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. Numbers & Letters EFFICIENCY module compares error detection to time. Greater "efficiency" defined as minimal errors during rapid processing. Slow, errorful processing is considered "inefficient". T scores indicate the degree to which processing efficiency differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores below 40 indicate decreased info processing efficiency. Scores above 60 indicate more efficient processing.
  T score with Mean=50, SD=10 | 41.0 (14.6)
Naming via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. Naming module measures language processing. Errorful naming is considered inefficient language processing. T scores indicate the degree to which language processing differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 47.6 (3.4)
List Learning List Immediate Recall via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. The List Learning List Immediate Recall module is one measure of short term memory. T scores indicate the degree to which short term memory differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 44.6 (2.4)
List Learning List Long Delayed Recall via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. The List Learning List Long Delayed Recall module is one measure of long term memory. T scores indicate the degree to which long term memory differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 44.6 (3.5)
Shape Learning Immediate Recognition via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. The Shape Learning Immediate Recognition module is another measure of short term memory. T scores indicate the degree to which short term memory differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 42.9 (3.0)
Shape Learning Delayed Recognition via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. The Shape Learning Delayed Recognition module is another measure of long term memory. T scores indicate the degree to which long term memory differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 41.3 (3.6)
Story Learning Phrase Unit Immediate Recall via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. The Story Learning Phrase Unit Immediate Recall module is another measure of short term memory. T scores indicate the degree to which short term memory differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 43.2 (2.9)
Story Learning Phrase Unit Delayed Recall via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. The Story Learning Phrase Unit Delayed Recall module is another measure of long term memory. T scores indicate the degree to which long term memory differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 43.7 (2.3)
Design Construction via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. Design Construction module is one measure of visuospatial processing. T scores indicate the degree to which visuospatial processing differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 41.4 (3.5)
Mazes via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. Mazes module is one measure of executive functioning. T scores indicate the degree to which executive functioning differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 39.8 (2.9)
Categories via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. Categories module is another measure of executive functioning. T scores indicate the degree to which executive functioning differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 41.8 (2.2)
Word Generation via Neuropsychological Assessment Battery [Mean (Standard Deviation); unit: T score with Mean=50, SD=10] — The Neuropsychological Assessment Battery is a comprehensive, demographically normalized battery of tests of neurocognitive function. The Word Generation module is another measure of executive functioning. T scores indicate the degree to which executive functioning differs from that of healthy demographically matched individuals. T-score of 50 is the mean. Scores significantly below 40 indicate decreased performance. Scores significantly above 60 indicate stronger ability compared to healthy demographically matched persons.
  T score with Mean=50, SD=10 | 45.0 (3.7)
Full Scale Intelligence Quotient (FSIQ) via Wechsler Test of Adult Reading [Mean (Standard Deviation); unit: units on a scale from 28 to 210] — The Wechsler Test of Adult Reading is a test of cognitive ability. The full scale intelligence quotient (FSIQ) estimate was obtained at Baseline to provide an estimate of premorbid cognitive functioning and to serve as a covariate for neurocognitive analyses. FSIQ population mean =100, SD = 15. By convention scores 130- 210 are very superior; 120-129 superior; 110-119 high average. Scores 90-109 are considered to be in the "average" range. Scores 80-89 are low average; 70-79 borderline; 28-69 are classified as extremely low.
  units on a scale from 28 to 210 | 95.8 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Radiation Necrosis and Cerebral Edema After a Single Treatment of Low Dose Intra-arterial Avastin (Bevacizumab)
Description: Imaging response to therapy will be quantitatively assessed on MRI using volumetric analysis. Regions of T2 and FLAIR prolongation above contralateral white matter will be calculated and quantified in cubic centimeters. Region of interest (ROI) will be created using a semi-automated, thresholding and region-growing technique. Enhancement of the lesion will be calculated using similar volumetric ROI analysis with a contrast threshold of 40% above background and measured in cubic centimeters.
Time Frame: Baseline (before treatment), and 3 months and 12 months after single dose intra-arterial Avastin (bevacizumab)
Population: 10 adult subjects presented with medically refractory radiation necrosis of the brain and disabling headache. All were treated with steroids prior to study enrollment.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Low-dose Intra-arterial Avastin (Bevacizumab)
Number analyzed (Participants) | 10
cm^3
  Vol EDEMA at Baseline | 86.8 (95.9)
  Vol EDEMA at 3 months | 38.6 (37.5)
  Vol EDEMA at 12 months: number analyzed (Participants) | 8
  Vol EDEMA at 12 months | 32.6 (33.7)
  Vol Radiation Necrosis at Baseline | 14.5 (12.1)
  Vol Radiation Necrosis at 3 months | 6.6 (7.5)
  Vol Radiation Necrosis at 12 months: number analyzed (Participants) | 8
  Vol Radiation Necrosis at 12 months | 3.2 (3.3)
Statistical Analysis 1: Comparison: Low-dose Intra-arterial Avastin (Bevacizumab); CHANGE IN VOLUME OF RADIATION NECROSIS: To explore durability of radiographic responses, we invoked a linear mixed model in which we addressed heterogeneity of time points by fitting the most appropriate model among compound symmetry, Huyhn-Felt structure, and an unstructured covariance matrix (multivariate analysis of variance); Test type: Other; p = 0.012, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; F(1,14) = 8.29; eta^2 = 0.37
Statistical Analysis 2: Comparison: Low-dose Intra-arterial Avastin (Bevacizumab); CHANGE IN VOLUME OF CEREBRAL EDEMA: To explore durability of radiographic responses, we invoked a linear mixed model in which we addressed heterogeneity of time points by fitting the most appropriate model among compound symmetry, Huyhn-Felt structure, and an unstructured covariance matrix (multivariate analysis of variance); Test type: Other; p = 0.09, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; F(1,14) = 3.29; eta^2 = 0.19

2. Secondary Outcome: Change in Headache Associated Morbidity Measured With MIDAS TOTAL SCORE After a Single Treatment of Low Dose Intra-arterial Avastin (Bevacizumab) Will be Measured.
Description: We will determine how severely headache affect the patient's life before and after treatment by performing the Migraine Disability Assessment (MIDAS) questionnaire. MIDAS TOTAL SCORE is the sum of Items 1 through 5. A Total Score of 0-5 signifies little or no disability, score of 6-10 signifies mild disability, score of 11-20 signifies moderate disability, and score of 21+ signifies severe disability. The theoretical maximum score would be 450.
Time Frame: Baseline (before treatment), and 6 weeks, 3 months, 6 months, 9 months, and 12 months after single dose intra-arterial Avastin (bevacizumab)
Population: 10 adult subjects presented with medically refractory radiation necrosis of the brain and disabling headache.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-dose Intra-arterial Avastin (Bevacizumab)
Number analyzed (Participants) | 10
score on a scale
  MIDAS TOTAL at Baseline | 81.7 (110.1)
  MIDAS TOTAL at 6 weeks | 49.7 (66.6)
  MIDAS TOTAL at 3 months | 22.1 (30.3)
  MIDAS TOTAL at 6 months | 28.3 (46.2)
  MIDAS TOTAL at 9 months | 24.4 (33.7)
  MIDAS TOTAL at 12 months | 15.6 (26.5)
Statistical Analysis 1: Comparison: Low-dose Intra-arterial Avastin (Bevacizumab); To explore durability of clinical response, Migraine Disability Assessment (MIDAS) TOTAL SCORES were analyzed using a linear mixed model in which we addressed heterogeneity of time points by fitting the most appropriate model among compound symmetry, Huyhn Felt structure, and an unstructured covariance matrix (multivariate analysis of variance); Test type: Other; p = 0.02, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; F(5,34) = 2.74; eta^2 = 0.29

3. Secondary Outcome: Change in Headache Associated Morbidity Measured With MIDAS DAYS of HEADACHE After a Single Treatment of Low Dose Intra-arterial Avastin (Bevacizumab) Will be Measured.
Description: We will determine how severely headache affect the patient's life before and after treatment by performing the Migraine Disability Assessment (MIDAS) questionnaire. MIDAS DAYS of HEADACHE is Item 6 of the questionnaire which sums total number of days the patient had headache symptoms over the past 3 months regardless of headache severity or resultant disability. Min score of 0 days is the best possible score. Max Score of 90 days is worse possible score, meaning the patient experienced headache pain every day over past 3 months.
Time Frame: as for outcome 2
Population: 10 adult subjects presented with medically refractory radiation necrosis of the brain and disabling headache.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Low-dose Intra-arterial Avastin (Bevacizumab)
Number analyzed (Participants) | 10
Days
  MIDAS DAYS of HEADACHE at Baseline | 33.3 (29.8)
  MIDAS DAYS of HEADACHE at 6 weeks | 25.8 (35.0)
  MIDAS DAYS of HEADACHE at 3 months | 9.0 (9.3)
  MIDAS DAYS of HEADACHE at 6 months | 14.6 (14.1)
  MIDAS DAYS of HEADACHE at 9 months | 12.4 (17.6)
  MIDAS DAYS of HEADACHE at 12 months | 11.5 (17.0)
Statistical Analysis 1: Comparison: Low-dose Intra-arterial Avastin (Bevacizumab); To explore durability of clinical response, Migraine Disability Assessment (MIDAS) DAYS OF HEADACHE were analyzed using a linear mixed model in which we addressed heterogeneity of time points by fitting the most appropriate model among compound symmetry, Huyhn Felt structure, and an unstructured covariance matrix (multivariate analysis of variance); Test type: Other; p = 0.019, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; F(5,34) = 3.17; eta^2 = 0.37

4. Secondary Outcome: Change in Headache Associated Morbidity Measured With MIDAS PAIN LEVEL After a Single Treatment of Low Dose Intra-arterial Avastin (Bevacizumab) Will be Measured.
Description: We will determine how severely headache affect the patient's life before and after treatment by performing the Migraine Disability Assessment (MIDAS) questionnaire. MIDAS PAIN LEVEL is Item 7 which rates the 3-month average headache PAIN LEVEL on scale from 0 to 10 where 0 = no pain at all, and 10 = pain as bad as it can be.
Time Frame: as for outcome 2
Population: 10 adult subjects presented with medically refractory radiation necrosis of the brain and disabling headache.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-dose Intra-arterial Avastin (Bevacizumab)
Number analyzed (Participants) | 10
score on a scale
  MIDAS PAIN LEVEL at Baseline | 6.9 (2.2)
  MIDAS PAIN LEVEL at 6 weeks | 6.4 (1.8)
  MIDAS PAIN LEVEL at 3 months | 4.7 (2.9)
  MIDAS PAIN LEVEL at 6 months | 5.0 (2.9)
  MIDAS PAIN LEVEL at 9 months | 4.8 (3.0)
  MIDAS PAIN LEVEL at 12 months | 4.8 (3.5)
Statistical Analysis 1: Comparison: Low-dose Intra-arterial Avastin (Bevacizumab); To explore durability of clinical response, Migraine Disability Assessment (MIDAS) MIDAS PAIN LEVEL data were analyzed using a linear mixed model in which we addressed heterogeneity of time points by fitting the most appropriate model among compound symmetry, Huyhn Felt structure, and an unstructured covariance matrix (multivariate analysis of variance); Test type: Other; p = 0.0006, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; F(5,35) = 3.96; eta^2 = 0.3

5. Secondary Outcome: Change in Headache Measured With Headache Impact Test (HIT-6) After a Single Treatment of Low Dose Intra-arterial Avastin (Bevacizumab)
Description: Quantitative change in headache will be assessed by performing the Headache Impact Test (HIT-6), which is a fixed-length 6-item questionnaire. The score for this questionnaire can range from 36 to 78, with 36 indicating minimum headache impact and the max score of 78 indicating worst possible headache impact.
Time Frame: as for outcome 2
Population: 10 adult subjects presented with medically refractory radiation necrosis of the brain and disabling headache. All 10 received single treatment of low dose intra-arterial bevacizumab.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-dose Intra-arterial Avastin (Bevacizumab)
Number analyzed (Participants) | 10
score on a scale
  Headache Impact Test-6, Baseline | 62.4 (7.5)
  Headache Impact Test-6, 6 Weeks | 54.5 (11.4)
  Headache Impact Test-6, 3 months | 52.3 (13.0)
  Headache Impact Test-6, 6 months | 53.3 (13.6)
  Headache Impact Test-6, 9 months | 53.2 (15.4)
  Headache Impact Test-6, 12 months: number analyzed (Participants) | 8
  Headache Impact Test-6, 12 months | 52.1 (14.4)
Statistical Analysis 1: Comparison: Low-dose Intra-arterial Avastin (Bevacizumab); To explore durability of clinical response, Headache Impact Test (HIT-6™) scores were analyzed using a linear mixed model in which we addressed heterogeneity of time points by fitting the most appropriate model among compound symmetry, Huyhn-Felt structure, and an unstructured covariance matrix (multivariate analysis of variance); Test type: Other; p = 0.02, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; F(5, 35) = 2.98; eta^2 = 0.30

6. Secondary Outcome: Change in Functional Status After a Single Treatment of Low Dose Intra-arterial Bevacizumab
Description: Quantitative change in functional status will be assessed by performing Karnofsky Performance Status Scale (KPS). The KPS score can range from 0 to 100 where 0 is dead and 100 is fully alive and normal with no complaints and no evidence of disease.
Time Frame: Baseline (before treatment), Day 1, and at 3 months, and 12 months after single dose intra-arterial Avastin (bevacizumab)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low-dose Intra-arterial Bevacizumab
Number analyzed (Participants) | 10
units on a scale
  Karnofsky at Baseline | 79.0 (9.9)
  Karnofsky at Day 1 | 81.0 (7.4)
  Karnofsky at Month 3 | 83.0 (11.6)
  Karnofsky at Month 12: number analyzed (Participants) | 8
  Karnofsky at Month 12 | 86.3 (7.4)
Statistical Analysis 1: Comparison: Low-dose Intra-arterial Bevacizumab; To explore durability of clinical response, Karnofsky Performance Status Scale (KPS) data were analyzed using a linear mixed model in which we addressed heterogeneity of time points by fitting the most appropriate model among compound symmetry, Huyhn-Felt structure, and an unstructured covariance matrix (multivariate analysis of variance); Test type: Other; p = 0.23, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; F(2,14) = 1.62; eta^2 = 0.19

7. Secondary Outcome: Change in Steroid Usage After a Single Treatment of Low Dose Intra-arterial Avastin (Bevacizumab)
Description: To assess the utility of intra-arterial (IA) bevacizumab treatment in allowing decreased steroid usage, total cumulative days of steroid usage were compared between the 12 months PRIOR TO and the 12 months IMMEDIATELY FOLLOWING IA bevacizumab. Days of steroid usage were tabulated via medical history and chart review at the baseline visit for the 12 months prior to IA bevacizumab and post-treatment on days 0 and 1, week 6, and months 3, 6, 9 and 12 for the 12 month total after IA bevacizumab treatment. Excluding topical steroid preparations, all days of enteral or parenteral steroid intake of any dose were included in the cumulative summation.
Time Frame: 12 months prior to single dose of IA bevacizumab; 12 months following single dose of IA bevacizumab
Population: 10 adult patients age 31.0 (IQR 24.3, 42.8) years, including 8 (80%) women, 2 (20%) men, 9 (90%) white, 1 (10%) black, 9 (90%) Non-Hispanic, and 1 (10%) Hispanic
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Low-dose Intra-arterial Avastin (Bevacizumab)
Number analyzed (Participants) | 10
Days
  12 months PRIOR to IA bevacizumab | 61.5 [0 to 156.25]
  12 months AFTER IA bevacizumab | 13.0 [0 to 87.25]
Statistical Analysis 1: Comparison: Low-dose Intra-arterial Avastin (Bevacizumab); Wilcoxon signed rank test (2-sided) was used to compare the total number of days on steroids in the 12 months prior versus the 12 months immediately following single dose IA Avastin (bevacizumab); Test type: Other; p = 0.374, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05; Z = -0.889; Pearson's r = -0.199

8. Secondary Outcome: Post-operative Neurocognitive Change After Intra-arterial Bevacizumab
Description: In order to investigate post-operative changes in Neurocognitive performance after intra-arterial bevacizumab, patients who consented underwent formal neuropsychological battery testing. Sixteen subtests from the Neuropsychological Assessment Battery (Stern & White, PAR Inc.) were chosen for brevity, sensitivity, and due to the wide range of available normative data (ages 18-97). For each subtest, T-score = 50 is the normative mean with SD = 10. Thus T-scores of 40-60 are within one standard deviation of the mean and are considered generally normal. Scores increasingly below 40 indicate decreased neurocognitive performance compared to healthy demographically matched persons. Scores significantly above 60 indicate increase neurocognitive performance compared to healthy demographically matched persons.
Time Frame: Baseline (before bevacizumab), and 3 months and 12 months after single dose intra-arterial Avastin (bevacizumab)
Population: 10 adult subjects, 2 male and 8 female, 1 black and 9 white, 1 Hispanic and 9 non-Hispanic, recruited from outpatient medical clinics at 2 academic medical centers (5 subjects per center) between Nov 2016 and Jan 2018. 2 subjects experienced progression of radiation necrosis requiring intervention at approx. month 11. Their 12-month data are not included in the Neurocognitive reporting.
Measure: Mean (Standard Deviation); unit: T score where mean T=50, SD=10
Arm/Group | Low-dose Intra-arterial Bevacizumab
Number analyzed (Participants) | 10
T score where mean T=50, SD=10
  Digits Forward at Baseline | 41.1 (11.8)
  Digits Forward at 3 months | 44.1 (12.2)
  Digits Forward at 12 months: number analyzed (Participants) | 8
  Digits Forward at 12 months | 42.3 (11.7)
  Digits Backward at Baseline | 44.9 (8.3)
  Digits Backward at 3 months | 44.9 (11.9)
  Digits Backward at 12 months: number analyzed (Participants) | 8
  Digits Backward at 12 months | 40.3 (13.1)
  Numbers & Letters SPEED at Baseline | 38.2 (10.7)
  Numbers & Letters SPEED at 3 months | 36.7 (10.8)
  Numbers & Letters SPEED at 12 months: number analyzed (Participants) | 8
  Numbers & Letters SPEED at 12 months | 36.8 (10.7)
  Numbers & Letters Errors at BASELINE | 44.6 (12.0)
  Numbers & Letters Errors at 3 months | 47.4 (12.6)
  Numbers & Letters Errors at 12 months: number analyzed (Participants) | 8
  Numbers & Letters Errors at 12 months | 52.9 (10.1)
  Numbers & Letters EFFICIENCY at Baseline | 41.0 (14.6)
  Numbers & Letters EFFICIENCY at 3 Months | 36.6 (11.8)
  Numbers & Letters EFFICIENCY at 12 months: number analyzed (Participants) | 8
  Numbers & Letters EFFICIENCY at 12 months | 36.6 (11.1)
  Naming at BASELINE | 47.6 (10.6)
  Naming at 3 months | 49.9 (7.3)
  Naming at 12 months: number analyzed (Participants) | 8
  Naming at 12 months | 49.1 (10.9)
  List Learning List Immediate Recall at BASELINE | 44.6 (7.7)
  List Learning List Immediate Recall at 3 months | 44.2 (13.1)
  List Learning List Immediate Recall at 12 months: number analyzed (Participants) | 8
  List Learning List Immediate Recall at 12 months | 46.4 (7.8)
  List Learning List Long Delayed Recall at BASELINE | 44.6 (11.1)
  List Learning List Long Delayed Recall at 3 months | 42.6 (11.0)
  List Learning List Long Delayed Recall at 12 months: number analyzed (Participants) | 8
  List Learning List Long Delayed Recall at 12 months | 51.3 (12.1)
  Shape Learning Immediate Recognition at BASELINE | 42.9 (9.5)
  Shape Learning Immediate Recognition at 3 months | 48.6 (10.7)
  Shape Learning Immediate Recognition at 12 months: number analyzed (Participants) | 8
  Shape Learning Immediate Recognition at 12 months | 50.0 (11.3)
  Shape Learning Delayed Recognition at BASELINE | 41.3 (11.3)
  Shape Learning Delayed Recognition at 3 months | 46.0 (12.2)
  Shape Learning Delayed Recognition at 12 months: number analyzed (Participants) | 8
  Shape Learning Delayed Recognition at 12 months | 47.3 (9.1)
  Story Learning Phrase Unit Immediate Recall at BASELINE | 43.2 (9.2)
  Story Learning Phrase Unit Immediate Recall at 3 months | 47.1 (12.7)
  Story Learning Phrase Unit Immediate Recall at 12 months: number analyzed (Participants) | 8
  Story Learning Phrase Unit Immediate Recall at 12 months | 49.6 (12.8)
  Story Learning Phrase Unit Delayed Recall at BASELINE | 43.7 (7.3)
  Story Learning Phrase Unit Delayed Recall at 3 months | 48.5 (9.2)
  Story Learning Phrase Unit Delayed Recall at 12 months: number analyzed (Participants) | 8
  Story Learning Phrase Unit Delayed Recall at 12 months | 47.1 (8.0)
  Design Construction at BASELINE | 41.4 (11.1)
  Design Construction at 3 months | 41.6 (14.3)
  Design Construction at 12 months: number analyzed (Participants) | 8
  Design Construction at 12 months | 45.8 (9.6)
  Mazes at BASELINE | 39.8 (9.2)
  Mazes at 3 months | 43.3 (12.3)
  Mazes at 12 months: number analyzed (Participants) | 8
  Mazes at 12 months | 43.0 (11.7)
  Categories at BASELINE | 41.8 (6.8)
  Categories at 3 months | 44.5 (10.4)
  Categories at 12 months: number analyzed (Participants) | 8
  Categories at 12 months | 39.9 (8.2)
  Word Generation at BASELINE | 45.0 (11.8)
  Word Generation at 3 months | 45.6 (9.8)
  Word Generation at 12 months: number analyzed (Participants) | 8
  Word Generation at 12 months | 49.0 (11.3)
Statistical Analysis 1: Comparison: Low-dose Intra-arterial Bevacizumab; DIGITS FORWARD: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the DIGITS FORWARD variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.660, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 0.451; partial eta^2 = 0.153
Statistical Analysis 2: Comparison: Low-dose Intra-arterial Bevacizumab; DIGITS BACKWARD: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the DIGITS BACKWARD variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.100, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 3.78; partial eta^2 = 0.602
Statistical Analysis 3: Comparison: Low-dose Intra-arterial Bevacizumab; NUMBERS & LETTERS SPEED: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the NUMBERS & LETTERS SPEED variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.149, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 2.847; partial eta^2 = 0.532
Statistical Analysis 4: Comparison: Low-dose Intra-arterial Bevacizumab; NUMBERS & LETTERS ERRORS: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the NUMBERS & LETTERS ERRORS variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.041, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 6.470; partial eta^2 = 0.721
Statistical Analysis 5: Comparison: Low-dose Intra-arterial Bevacizumab; NUMBERS & LETTERS EFFICIENCY: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the NUMBERS & LETTERS EFFICIENCY variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.124, One way Repeat Meas ANOVA; F (2,5) = 3.256; partial eta^2 = 0.566
Statistical Analysis 6: Comparison: Low-dose Intra-arterial Bevacizumab; NAMING: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the NAMING variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.898, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 0.110; partial eta^2 = 0.042
Statistical Analysis 7: Comparison: Low-dose Intra-arterial Bevacizumab; LIST LEARNING LIST IMMEDIATE RECALL: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the LIST LEARNING LIST IMMEDIATE RECALL variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.754, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 0.299; partial eta^2 = 0.107
Statistical Analysis 8: Comparison: Low-dose Intra-arterial Bevacizumab; LIST LEARNING LIST LONG DELAYED RECALL: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the LIST LEARNING LIST LONG DELAYED RECALL variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.031, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 7.556; partial eta^2 = 0.751
Statistical Analysis 9: Comparison: Low-dose Intra-arterial Bevacizumab; SHAPE LEARNING IMMEDIATE RECOGNITION: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the SHAPE LEARNING IMMEDIATE RECOGNITION variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.426, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 1.018; partial eta^2 = 0.289
Statistical Analysis 10: Comparison: Low-dose Intra-arterial Bevacizumab; SHAPE LEARNING DELAYED RECOGNITION: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the SHAPE LEARNING DELAYED RECOGNITION variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.326, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 1.412; partial eta^2 = 0.361
Statistical Analysis 11: Comparison: Low-dose Intra-arterial Bevacizumab; STORY LEARNING PHRASE UNIT IMMEDIATE RECALL: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the STORY LEARNING PHRASE UNIT IMMEDIATE RECALL variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.790, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 0.247; partial eta^2 = 0.090
Statistical Analysis 12: Comparison: Low-dose Intra-arterial Bevacizumab; STORY LEARNING PHRASE UNIT DELAYED RECALL: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the STORY LEARNING PHRASE UNIT DELAYED RECALL variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.505, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 0.786; partial eta^2 = 0.239
Statistical Analysis 13: Comparison: Low-dose Intra-arterial Bevacizumab; DESIGN CONSTRUCTION: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the DESIGN CONSTRUCTION variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.080, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 4.362; partial eta^2 = 0.636
Statistical Analysis 14: Comparison: Low-dose Intra-arterial Bevacizumab; MAZES: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the MAZES variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.052, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 5.654; partial eta^2 = 0.693
Statistical Analysis 15: Comparison: Low-dose Intra-arterial Bevacizumab; CATEGORIES: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the CATEGORIES variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.968, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 0.033; partial eta^2 = 0.013
Statistical Analysis 16: Comparison: Low-dose Intra-arterial Bevacizumab; WORD GENERATION: To explore post-operative change in Neurocognitive performance after intra-arterial bevacizumab, repeated measures ANOVA was performed for the WORD GENERATION variable across 3 time points (BL, 3 months, 12 months) where IQ was placed in the model as covariate; Test type: Other; p = 0.469, One way Repeat Meas ANOVA — The threshold for statistical significance was p < 0.05; F(2,5) = 0.884; partial eta^2 = 0.261

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse Event Monitoring performed on Day 0, Day 1, Week 6, Month 3, and Month 12
Arm/Group | Low-dose Intra-arterial Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Intra-arterial Bevacizumab (N=10)
Seizure (Nervous system disorders) | 2 (2) — Month 6 Pt 20 min non-responsive but appeared awake. Ambulance. Brain MRI decr edema no acute infarct or hemorrh. D/C home. Another Pt month 6 seizure activity w dizziness, chest pain, left jaw pain and left arm pain and numbness, double vision
Acute encephalopathy (Nervous system disorders) | 1 (1) — Pt admitted month 9 for 1-Confusion 2-Intermittent diaphoresis 3-Heat/cold intolerance 4-Mild abd Pain 5-Vomiting 6-Unsteadiness. Brain CT/MRI no sig change target area, age related ischemic changes. Workup neg. Meds held pt improved D/Ced home.
Double Vision (Nervous system disorders) | 1 (1) — Double vision on Day 1 with dizziness reported after transferred into TCU per protocol. Investigator notified, patient transferred to ICU, symptoms resolved 2 hours after onset.
Chest Pain (Cardiac disorders) | 1 (1) — Pt has history of chest pain but symptoms worsened and were associated with Month 6 episode of seizures
Headache (Nervous system disorders) | 1 (1) — Month 9 Pt having recurrent worsening headaches, Brain MRI showed peri-lesion radiation necrosis with residual AVM. Pt opted for surgical resection of simple supra-tentorial AVM and Radiation necrosis in the Perisylvian and insular region.
Dizziness (Nervous system disorders) | 1 (1) — Day 1 Double vision with dizziness reported after transferred into TCU per protocol. Investigator notified, patient transferred to ICU, symptoms resolved 2 hours after onset.
Dysarthria (Nervous system disorders) | 1 (1) — Day 1 Pt developed acute onset Dysarthria followed by Lt. UE and LE Hemiparesis. Evaluated in ED, Brain CT/MRI and EEG revealed no sig changes, Hospitalized x 8 d started on steroids and Keppra (for poss seizure) weakness improved to LUE 5/5, LLE 3/5
Left Lower Extremity Hemiparesis (Nervous system disorders) | 1 (1) — Day 1 Pt developed acute onset Dysarthria followed by Lt. UE and LE Hemiparesis. Evaluated in ED, Brain CT/MRI and EEG revealed no sig changes, Hospitalized x 8 d started on steroids and Keppra (for poss seizure) weakness improved to LUE 5/5, LLE 3/5
Left Upper Extremity Hemiparesis (Nervous system disorders) | 1 (1) — Day 1 Pt developed acute onset Dysarthria followed by Lt. UE and LE Hemiparesis. Evaluated in ED, Brain CT/MRI and EEG revealed no sig changes, Hospitalized x 8 d started on steroids and Keppra (for poss seizure) weakness improved to LUE 5/5, LLE 3/5
Cerebral Edema (Nervous system disorders) | 1 (1) — Month 8 Pt having symptoms of cerebral edema, Brain MRI showed interval increase in edema and radiation necrosis. Pt opted for 2 cycles of IV Avastin with subsequent improvement in symptoms and MRI findings.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Intra-arterial Bevacizumab (N=10)
1st degree AV block (Cardiac disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) — Acne Related to Decadron
Altered Mental Status (Nervous system disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Anxiety (Nervous system disorders) | 1 (1)
Asthma episode (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilateral lower leg edema (Vascular disorders) | 1 (1)
Blurred vision (Eye disorders) | 4 (6)
Cervical strain (Musculoskeletal and connective tissue disorders) | 1 (1) — Cervical strain due to MVA
Confusion (Nervous system disorders) | 1 (2)
Decreased appetite (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Expressive aphasia (Nervous system disorders) | 1 (1)
Fall (General disorders) | 2 (2)
Fracture Left Hand (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 5 (7) — 1 episode Frontal Headache from MVA; 1 episode Headache; 1 episode Right sided headache; 1 episode Headaches with vertigo; 3 episodes worsening headache
Generalized Anxiety (Psychiatric disorders) | 1 (1)
Generalized Malaise (General disorders) | 1 (1)
hair loss (Skin and subcutaneous tissue disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Head Trauma (Injury, poisoning and procedural complications) | 1 (1)
Hypercholesterolemia (General disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Hypertriglyceridemia (General disorders) | 1 (1)
Inability to focus (Eye disorders) | 1 (1)
Inability to focus attention (Nervous system disorders) | 1 (1)
Incomplete Spontaneous Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) — Increased dizziness
Eye twitches (Eye disorders) | 1 (1) — Left eye twitches
Homonymous Hemianopia (Eye disorders) | 1 (1) — Left Homonymous Hemianopia
Leg skin tear non-healing wound (Skin and subcutaneous tissue disorders) | 1 (1) — Left Leg skin tear non-healing wound
Leg traumatic injury (Injury, poisoning and procedural complications) | 1 (1) — Left leg traumatic injury
Loss of appetite (Gastrointestinal disorders) | 1 (1)
Loss of vision (Eye disorders) | 1 (1) — loss of vision X 30 seconds
Lower Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Major Depressive Disorder (Psychiatric disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — Mild Abdominal Pain
Nausea (Gastrointestinal disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nosebleeds (General disorders) | 1 (1)
Panic attacks (Psychiatric disorders) | 1 (1)
Personality Changes (Psychiatric disorders) | 1 (1) — Personality Changes including anger
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Numbness (Nervous system disorders) | 2 (2) — 1 episode Intermittent Numbness in the bottom; 1 episode Whole body numbness
Scalp Pain (Skin and subcutaneous tissue disorders) | 1 (1) — Left vertex scalp soreness
Ankle sprain due to fall (Injury, poisoning and procedural complications) | 1 (2) — Right ankle sprain due to fall
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Right Hip Radiating Pain
Inner Ear pain (Ear and labyrinth disorders) | 1 (1) — Right Inner Ear pain
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) — right knee pain from MVA
Cold sensation leg (Nervous system disorders) | 1 (1) — Right leg cold sensation knee to foot
Leg cramps (Musculoskeletal and connective tissue disorders) | 2 (3)
Leg Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1) — Right Leg Muscle aches
Partial toenail ingrown (Musculoskeletal and connective tissue disorders) | 1 (1) — Right partial toenail ingrown
Calf muscle loss of tone (Nervous system disorders) | 1 (1) — Rt Calf muscle loss of tone
Seizures (Nervous system disorders) | 2 (2)
Generalized Seizures (Nervous system disorders) | 1 (1)
Tonic/clonic Seizures (Nervous system disorders) | 1 (2)
Shot term memory problems (Nervous system disorders) | 1 (1)
Steroid Induced Hyperglycemia (Endocrine disorders) | 1 (1)
Vision loss in left eye (Eye disorders) | 1 (1) — temporary vision loss in left eye
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Traumatic Fall (Injury, poisoning and procedural complications) | 2 (2)
Trouble performing simple tasks (Nervous system disorders) | 1 (1)
Unsteadiness (Nervous system disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Visual seizure (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight Loss (Metabolism and nutrition disorders) | 1 (1)
Whole body shaking associated with seizures (Nervous system disorders) | 1 (1)
Worsening Acne on extremities (Skin and subcutaneous tissue disorders) | 1 (1)
Worsening chest pain (Cardiac disorders) | 1 (1)
Worsening of left sided weakness (Nervous system disorders) | 1 (1)
Worsening of striae bilateral arms (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Pilot Phase 2 Single Arm Clinical Trial with small number of patients. Not powered sufficiently to provide definitive proof for change in current standard of care of medically refractory radiation necrosis of the brain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT02819479/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT02819479/ICF_001.pdf